CLINICAL TRIAL: NCT03103373
Title: Assessment of Plasma Lactate in Patients Underwent Non-cardiac Surgery Monitoring by Transthoracic Echocardiography
Brief Title: Assessment of Plasma Lactate in Non-cardiac Surgery Monitoring by Transthoracic Echocardiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Marcello F Salgado Filho, MD, Professor of Anesthesiology, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 60721816.9.0000.5139
Record Dates: First submitted 2017-03-10; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia
Keywords: Echocardiography; anesthesia; general surgery
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: The study is a clinical trial, prospective and random type, in which 60 patients, of both genders, aged between 18 and 80 years, who will undergo major abdominal surgery, divided in two groups.
  Patients will be randomly divided into two groups with 35 patients:
  Conventional Group, Transthoracic Echocardiogram Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional monitor group (Active Comparator): Patients will be monitoring with invasive blood pressure, central venus catheter, plasma lactate, urinary output, oximeter, capnography and electrocardiography Echocardiography group: Patients will be monitoring with echocardiography, invasive blood pressure, central venus catheter, plasma lactate, urinary output, oximeter, capnogrphy and electrocardiography
  Interventions: Device: Conventional monitor
- Echocardiography group (Active Comparator): Patients will be monitoring with echocardiography, invasive blood pressure, central venus catheter, plasma lactate, urinary output, oximeter, capnography and electrocardiography
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Conventional monitor — Patients underwent non-cardiac surgery will be monitoring by regular monitors
  Arms: Conventional monitor group
Device: Echocardiography — Patients will be monitoring by regular monitors plus echocardiography
  Arms: Echocardiography group

SUMMARY:
The study is a clinical trial, prospective and randomized of 60 patients of both genders, aged between 18 and 80 years, underwent major abdominal surgery. This study aims to compare plasma lactate levels in patients underwent major abdominal surgery (colectomy, gastrectomy, esophagectomy, pancreatectomy, Wertheim Meigs, liver and spleen surgeries) monitored by echocardiography or by conventional techniques (mean arterial pressure , Central venous pressure).

DETAILED DESCRIPTION:
The study is a clinical trial, prospective and randomized of 60 patients of both genders, aged between 18 and 80 years, underwent major abdominal surgery. This study aims to compare plasma lactate levels in patients underwent major abdominal surgery (colectomy, gastrectomy, esophagectomy, pancreatectomy, Wertheim Meigs, liver and spleen surgeries) monitored by echocardiography or by conventional techniques (mean arterial pressure , Central venous pressure).

The investigators expect to observe a decrease in plasma lactate levels in patients submitted to echocardiographic monitoring when compared to patients submitted to conventional monitoring. In this way, to demonstrate that the routine use of transthoracic echocardiography in patients submitted to large surgery improves the clinical outcomes of these patients and presents a lower hospital cost.

The surgical indication will obey the criteria of the Federal University of Juiz de Fora surgery service, after clinical examination and routine preoperative laboratory tests (complete blood count, complete coagulogram, plasma sodium, potassium Plasma urea and plasma creatinine, blood glucose and liver function test), resting electrocardiogram and chest X-ray. All patients who agree to participate in the study will sign an Informed Consent Term in the preanesthetic evaluation (Appendix 1).

Patients will be computer randomly form by the GraphPad Prisma® program into two groups with 30 patients:

Conventional Group, Transthoracic Echocardiogram Group, All survey data will be noted in the Protocol Data Sheet (Appendix 2). Patients will be anesthetized by the researcher Dr. Marcello Fonseca Salgado Filho, who will also be responsible for performing the intraoperative TTE examination.

ELIGIBILITY:
Inclusion Criteria:

ages between 18 and 80 years.

* both genders
* Large abdominal surgeries
* Elective surgeries

Exclusion Criteria:

* Emergency surgeries

  * Surgeries of the abdominal aorta
  * Ejection fraction <30%
  * Blood creatinine levels> 2.0mg / dl
  * Glycemia> 200 g / dl
  * Do not agree to participate in the study
  * Bowel obstruction
  * Sepsis
  * Bilirubin> 300 g / dl
  * Alcoholism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
plasma lactate | 10 minutes after intubation, before incision
  The plasma lactate will be collected in the arterial line
plasma lactate | 10 min after the end of the surgery
  The plasma lactate will be collected in the arterial line

SECONDARY OUTCOMES:
Assessment heart rate | 10 minutes after intubation, before incision
  Heart rate
Assessment heart rate | 10 min after the end of the surgery
  Heart rate
Assessment blood pressure | 10 minutes after intubation, before incision
  blood pressure
Assessment blood pressure | 10 min after the end of the surgery
  blood pressure
Assessment venus oximetry | 10 minutes after intubation, before incision
  venus oximetry
Assessment venus oximetry | 10 min after the end of the surgery
  venus oximetry
Assessment arterial PH | 10 minutes after intubation, before incision
  arterial PH
Assessment arterial PH | 10 min after the end of the surgery
  arterial PH
Assessment fluid infusion | 10 min after the end of the surgery
  fluid infusion
Infection | 30 days after surgery
  Assessment sepsis
Surgery complications | 30 days after surgery
  Assessment fistulae
Post-operative mortality | 30 days after surgery
  death after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marcello F Salgado Filho, PhD, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Result] Lobo SM, Rezende E, Knibel MF, Silva NB, Paramo JA, Nacul FE, Mendes CL, Assuncao M, Costa RC, Grion CC, Pinto SF, Mello PM, Maia MO, Duarte PA, Gutierrez F, Silva JM Jr, Lopes MR, Cordeiro JA, Mellot C. Early determinants of death due to multiple organ failure after noncardiac surgery in high-risk patients. Anesth Analg. 2011 Apr;112(4):877-83. doi: 10.1213/ANE.0b013e3181e2bf8e. Epub 2010 Jun 8. PMID 20530615
- [Result] Grocott MP, Dushianthan A, Hamilton MA, Mythen MG, Harrison D, Rowan K; Optimisation Systematic Review Steering Group. Perioperative increase in global blood flow to explicit defined goals and outcomes following surgery. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD004082. doi: 10.1002/14651858.CD004082.pub5. PMID 23152223
- See also: anesthesia and analgesia — http://journals.lww.com/anesthesia-analgesia
- See also: cochrane — http://www.cochrane.org